CLINICAL TRIAL: NCT02820194
Title: A Randomized Phase III Trial on Stereotactic Body Radiation Therapy (SBRT) Versus Microwave Ablation (MWA) for Inoperable Colorectal Liver Metastases (CLM)
Brief Title: A Trial on SBRT Versus MWA for Inoperable Colorectal Liver Metastases (CLM)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not sufficient patient recruited
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, Medical Doctor, Istituto Clinico Humanitas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1559
Record Dates: First submitted 2016-06-24; First posted 2016-06-30 (Estimated); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Secondary Malignant Neoplasm of Liver
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stereotactic body radiation therapy (Active Comparator): Patients are treated with Stereotactic Body Radiation Therapy, a methodology for delivering a conformal high dose of radiation to the tumor and a minimal dose to surrounding critical tissues, with a hypofractionation schedule.
  Interventions: Radiation: Stereotactic Body Radiation Therapy
- Microwave Ablation (Active Comparator): Patients are treated with Microwave Ablation,a newer technology that utilizes high-frequency electromagnetic radiation to create thermal damage and coagulation necrosis.
  Interventions: Procedure: Microwave Ablation

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — Stereotactic body radiation is a therapy for delivering a conformal high dose of radiation to the tumor and a minimal dose to surrounding critical tissues, with a hypofractionation schedule
  Arms: Stereotactic body radiation therapy
Procedure: Microwave Ablation — Microwave ablation (MWA) is a newer technology that utilizes high-frequency electromagnetic radiation to create thermal damage and coagulation necrosis
  Arms: Microwave Ablation

SUMMARY:
The trial is designed to perform a rigorous evaluation of efficacy and tolerability of SBRT by means of a randomised, controlled trial in patients affected by inoperable colorectal liver metastases. The chosen comparator is MWA.

The two modality treatments (SBRT versus MWA) will be evaluated for short- and longer-term outcomes.

DETAILED DESCRIPTION:
The trial is a monocentric prospective, randomised controlled, unblinded, parallel-group superiority trial of Stereotactic Body Radiation Therapy (SBRT) versus Microwave Ablation (MWA) for the curative treatment of inoperable colorectal liver metastases. Patients will be randomised on an equal basis to either SBRT or MWA. The two modality treatments (SBRT versus MWA) will be evaluated for short- and longer-term outcomes. The key short-term outcomes will include assessment of local response rate and acute toxicity. Longer-term outcomes will concentrate on oncological aspects of the disease with analysis of disease-free and overall survival and local recurrence rates at 3-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Karnofsky index >70%
* Histological proven adenocarcinoma of the colon or rectum with radiological (by CT- or MRI) or histological-/cytological verified liver metastases.
* Metastases must be visible on diagnostic- and dose planning CT scans and on ultrasonography.
* The patient should not be suitable for surgical resection due to technical or patient-related conditions. Resectability must be judged by a trained hepatobiliary surgeon and discussed in a multidisciplinary team meeting.
* Presence of 1-3 lesions .
* Diameter ≤ 40 mm.
* All tumors should be feasible for treatment with each of the two modalities, SBRT and MWA
* Adequate liver function: bilirubin <1.5 mg/dl, alb> 3.5g/dl, normal PT/PTT except if the patient uses anticoagulants, liver enzymes<3 times upper limit of normal. No ascites.
* Renal function must be adequate for infusion of iv. contrast for CT-scan.
* Adequate bone marrow function: Hbg³8 g/dl, platelets³100.000 and leucocytes ³2.000/ml.
* Informed consent.
* Extrahepatic disease stable or in response after CT
* No previous abdominal radiation therapy (RT)

Exclusion Criteria:

* Uncontrolled primary tumor or extrahepatic disease
* Previous abdominal radiation therapy (RT) or other local conservative treatment on lesion target.
* Pregnant or breastfeeding patients.
* Prior malignancy within the last five years (except adequately treated basal cell carcinoma of the skin or in situ carcinoma of the skin or in situ carcinoma of the cervix, surgically cured, or localized prostate cancer without evidence of biochemical progression).
* Previous inclusion in this study.
* Underlying liver cirrhosis (Child-Pugh grade B or C).
* Ascites and/or relevant intra-hepatic biliary tract dilatation.
* Mental conditions rendering the patient incapable to understand the nature, scope, and consequences of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-06; Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Control of local disease | 18 months
  Evaluation of proportion of patients free from progression from starting radiotherapy

SECONDARY OUTCOMES:
Progression free-survival of treated patients | 18 months
  Evaluation of proportion of patients alive and free from progression
Overall survival of treated patients | 18 months
  Evaluation of proportion of patients alive
Incidence of acute and late complications | 18 months
  Evaluation of early and late post treatment complications

CONTACTS AND LOCATIONS:
Overall Officials: Marta Scorsetti, MD, Principal Investigator — Humanitas Cancer Center
Locations (1):
- Humanitas Research Hospital, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No